CLINICAL TRIAL: NCT03425253
Title: A Prospective, Open-label Study to Evaluate Sequential Treatment With BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine for Overall Improvement in Jawline Contour
Brief Title: Sequential Treatment With BELKYRA® Then Juvéderm® VOLUMA™ With Lidocaine for Overall Improvement in Jawline Contour
Acronym: JAWLINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO-MA-FAS-0513
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Contour
Keywords: Lower Face Contouring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BELKYRA® and Juvéderm® VOLUMA™ with Lidocaine (Experimental): BELKYRA® was injected into subcutaneous preplatysma fat tissue in the submental area (at least 1 plus up to 5 optional treatments, for maximum of 6 treatments 8 weeks apart). When the investigator and participant agreed that no further intervention was required to achieve the desired result, participants were eligible to receive VOLUMA™ treatment. VOLUMA™ was injected along the mandibular border, with an optional touch-up visit 2 weeks later if applicable.
  Interventions: Drug: BELKYRA®; Device: Juvéderm® VOLUMA™ with Lidocaine

INTERVENTIONS:
Drug: BELKYRA® — BELKYRA® was injected into preplatysma fat tissue in the submental area (at least 1 plus up to 5 optional treatments, for maximum of 6 treatments 8 weeks apart).
Device: Juvéderm® VOLUMA™ with Lidocaine — Juvéderm® VOLUMA™ with Lidocaine VOLUMA™ was injected along the mandibular border.

SUMMARY:
This study has been designed to evaluate the safety and effectiveness of sequential treatment with BELKYRA® (for the treatment of convexity and fullness associated with submental fat) and VOLUMA™ (to restore volume along the mandibular border) to enhance the overall contour of the jawline.

DETAILED DESCRIPTION:
Participants may be treated with up to 6 treatments with Belkyra, followed by treatment with Voluma. Participants will have opportunity to participation in a skin biopsy sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2 or above on Allergan Loss of Jawline Definition Scale (ALJDS)
* Grade 2 or 3 on reported Clinician-Rated Submental Fat Rating Scale (CR-SMFRS)
* Stable body weight for at least 26 weeks
* Accept the obligation to forego any treatment or behavior (e.g., unshaven facial hair; significant changes to dietary or exercise habits) during the participants participation in the study that may affect the assessments of the submental area

Exclusion Criteria:

* Grade 4 on Submental Skin Laxity Grade (SMSLG)
* Grade 4 on Allergan Jowl Fat Rating Scale (AJFRS)
* Body mass index (BMI) >35 kg/m^2
* History of, or current symptoms of dysphagia
* History of temporary, semi-permanent or permanent facial or neck dermal filler injections below the medial canthi at any time prior to treatment, or within 52 weeks before Screening for treatment above the medial canthi
* History of facial and/or neck plastic surgery, tissue grafting or permanent facial implants anywhere in the face or neck
* History of any intervention (e.g., liposuction, surgery, or lipolytic agents) to treat submental fat (SMF)
* Evidence of any cause of enlargement in the submental area other than localized SMF
* History of mesotherapy or ablative procedures to the face and/or neck 52 weeks before Screening
* History of skin resurfacing in the neck or submental area within 26 weeks before Screening
* Treatment with botulinum toxin injections in the neck or submental area within 26 weeks before Screening
* Participants on prescription topical retinoid therapy and/or topical hormone cream applied to the face, who have not been on a consistent dose regimen for at least 26 weeks before Screening and who are unable to maintain regimen for the study
* Systemic retinoid therapy within 52 weeks before Screening
* Current use of oral corticosteroids
* Is on a regimen of anticoagulation therapy (eg, warfarin, clopidogrel)
* Has current injection site inflammatory or infectious processes, abscess, an unhealed wound, or a known cancerous or precancerous lesion in chin, masseter, or submental region
* Planned oral surgery or other dental procedures (e.g., tooth extraction, orthodontia, or implantation) within 2 weeks prior to and after VOLUMA™ treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silberberg, Study Director — Allergan
Locations (3):
- Australia (3):
  - Darlinghurst Dermatology, Darlinghurst, New South Wales
  - Living Art, East Melbourne, Victoria
  - Dermatology Institute of Victoria, South Yarra, Victoria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants participated in the study at 3 study sites in Australia from 02 February 2018 to 05 December 2019.
Period: Overall Study
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Started | 58
Safety Analysis Set (Safety Analysis Set included participants who are defined as Full Analysis Set (FAS) participants and those participants who underwent biopsy procedure but did not receive the BELKYRA® treatment.) | 53
FAS (FAS population included all participants who received BELKYRA®.) | 53
Evaluable Set (ES) (ES population included all participants who received BELKYRA® plus VOLUMA™.) | 42
Completed | 42
Not Completed | 16
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 3
Not completed — Withdrew Consent | 6
Not completed — Did not Meet all Eligibility Criteria Defined in the Protocol | 5

BASELINE CHARACTERISTICS:
Population: FAS included all participants who received BELKYRA®.
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 51
  Race: Asian /Oriental | 1
  Race: Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Showed ≥ 1-point Jawline Improvement From Baseline on the Allergan Loss of Jawline Definition Scale (ALJDS), as Assessed by the Investigator
Description: The ALJDS was an investigator assessment of loss of jawline definition measured by a 5-point scale where: 0=none, 1=mild, 2=moderate, 3=severe, 4=extreme. Data is reported for both sides of the face, right side of the face and left side of the face.
Time Frame: Baseline (Day 0) to Week 58
Population: Evaluable Set (ES) included participants who received both study treatments (i.e., both BELKYRA® and VOLUMA™) and had a post-treatment efficacy assessment at the Exit Visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 42
percentage of participants
  Both Sides of the Face | 92.9 [80.5 to 98.5]
  Right Side of the Face | 92.9 [80.5 to 98.5]
  Left Side of the Face | 92.9 [80.5 to 98.5]

2. Secondary Outcome: Mean Change From Baseline to Last BELKYRA® Treatment on the ALJDS
Description: The ALJDS was an investigator and independent reviewer assessment of jawline contour measured by a 5-point scale where: 0=none, 1=mild, 2=moderate, 3=severe, 4=extreme. A negative change from baseline indicated improvement. The data is reported for both sides of the face, right side of the face and left side of the face.
Time Frame: Baseline (Day 0) to Last Treatment (Up to Week 48)
Population: FAS included all participants who received BELKYRA®. Number analyzed is the number of participants with available data at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine: BELKYRA® was injected into subcutaneous preplatysma fat tissue in the submental area (at least 1 plus up to 5 optional treatments, for maximum of 6 treatments 8 weeks apart).
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 53
score on a scale
  Investigator: Both Sides of Face, Baseline | 2.7 (0.52)
  Investigator: Both Sides of Face, Last Treatment | -0.6 (0.71)
  Investigator: Right Side of Face, Baseline | 2.5 (0.50)
  Investigator: Right Side of Face, Last Treatment | -0.6 (0.62)
  Investigator: Left Side of Face, Baseline | 2.6 (0.52)
  Investigator: Left Side of Face, Last Treatment | -0.6 (0.72)
  Independent Reviewer: Both Sides of Face, Baseline: number analyzed (Participants) | 51
  Independent Reviewer: Both Sides of Face, Baseline | 2.9 (1.04)
  Independent Reviewer: Both Sides of Face, Last Treatment: number analyzed (Participants) | 51
  Independent Reviewer: Both Sides of Face, Last Treatment | -0.3 (0.98)
  Independent Reviewer: Right Side of Face, Baseline: number analyzed (Participants) | 51
  Independent Reviewer: Right Side of Face, Baseline | 2.7 (1.10)
  Independent Reviewer: Right Side of Face, Last Treatment: number analyzed (Participants) | 51
  Independent Reviewer: Right Side of Face, Last Treatment | -0.1 (1.13)
  Independent Reviewer: Left Side of Face, Baseline: number analyzed (Participants) | 51
  Independent Reviewer: Left Side of Face, Baseline | 2.7 (1.03)
  Independent Reviewer: Left Side of Face, Last Treatment: number analyzed (Participants) | 51
  Independent Reviewer: Left Side of Face, Last Treatment | -0.4 (1.01)
Statistical Analysis 1: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Investigator: Both Sides of Face, Last Treatment; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference
Statistical Analysis 2: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Investigator: Right Side of Face, Last Treatment; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference
Statistical Analysis 3: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Investigator: Left Side of Face, Last Treatment; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference
Statistical Analysis 4: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Independent Reviewer: Both Sides of Face, Last Treatment; Test type: Other; p = 0.018, Paired t-test — P-value was based on paired t-test for the mean difference
Statistical Analysis 5: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Independent Reviewer: Right Side of Face, Last Treatment; Test type: Other; p = 0.301, Paired t-test — P-value was based on paired t-test for the mean difference
Statistical Analysis 6: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Independent Reviewer: Left Side of Face, Last Treatment; Test type: Other; p = 0.011, Paired t-test — P-value was based on paired t-test for the mean difference

3. Secondary Outcome: Mean Change From Baseline to Final Study Visit in the FACE-Q™ Satisfaction With Lower Face and Jawline Score
Description: The participant assessed satisfaction using the 5 items on the Satisfaction of Lower Face and Jawline module of the FACE-Q™ questionnaire, measured on a 4-point scale where: 1=very dissatisfied, 2=somewhat dissatisfied, 3=somewhat satisfied, 4=very satisfied. The Rasch transformed scale total score was 0 (worst) to 100 (best). A positive change from baseline indicated improvement.
Time Frame: Baseline (Day 0) to Week 58
Population: ES included participants who received both study treatments (i.e., both BELKYRA® and VOLUMA™) and had a post-treatment efficacy assessment at the Exit Visit.
Measure: Mean (Standard Deviation); unit: score on a score
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 42
score on a score
  Baseline | 24.1 (16.78)
  Change From Baseline to Week 58 | 55.9 (21.78)
Statistical Analysis 1: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference

4. Secondary Outcome: Mean Change From Baseline to Final Study Visit in the FACE-Q™ Appraisal of Neck
Description: The participant assessed satisfaction using the 10 items on the Appraisal of Neck module of the FACE-Q™ questionnaire measured on a 4-point scale where: 1=not at all, 2=a little, 3=moderately, 4=extremely. The Rasch transformed scale total score was 0 (worst) to 100 (best). A positive change from baseline indicated improvement.
Time Frame: Baseline (Day 0) to Week 58
Population: ES included participants who received both study treatments (i.e., both BELKYRA® and VOLUMA™) and had a post-treatment efficacy assessment at the Exit Visit. Overall number analyzed is the number of participants with available data at given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 30
score on a scale
  Baseline | 13.8 (8.85)
  Change From Baseline to Week 58: number analyzed (Participants) | 2
  Change From Baseline to Week 58 | -11.0 (13.44)
Statistical Analysis 1: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Test type: Other; p = 0.597, Paired t-test — P-value was based on paired t-test for the mean difference

5. Secondary Outcome: Mean Change From Baseline to Final Study Visit for FACE-Q™ Appraisal of Area Under Chin
Description: The participant assessed satisfaction using the 5 items on the Appraisal of Area Under Chin module of the FACE-Q™ questionnaire measured on a 4-point scale where: 1=not at all, 2=a little, 3=moderately, 4=extremely. The Rasch transformed scale total score was 0 (worst) to 100 (best). A negative change from baseline indicated worsening.
Time Frame: Baseline (Day 0) to Week 58
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 42
score on a scale
  Baseline | 60.1 (23.86)
  Change From Baseline to Week 58 | -45.4 (17.09)
Statistical Analysis 1: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference

6. Secondary Outcome: Mean Change From Baseline to Final Study Visit for Clinician-Reported Submental Fat Rating Scale (CR-SMFRS)
Description: The CR-SMFRS score was based on the investigator's clinical evaluation of the participant, where submental fullness was scored on a 5-point scale where: 0=absent, 1=mild, 2=moderate, 3=severe, and 4=extreme. A negative change from baseline indicated improvement.
Time Frame: Baseline (Day 0) to Week 58
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 42
score on a scale
  Baseline | 2.5 (0.50)
  Change From Baseline to Week 58 | -1.9 (0.67)
Statistical Analysis 1: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference

7. Secondary Outcome: Mean Change From Baseline to Final Study Visit for Patient-Reported Submental Fat Rating Scale (PR-SMFRS)
Description: The PR-SMFRS was based on the participant's response to the question "How much fat do you have under your chin right now?" and answered on a 5-point ordinal scale where: 0=no chin fat at all, 1=a slight amount of chin fat, 2=a moderate amount of chin fat, 3=a large amount of chin fat, and 4=a very large amount of chin fat. A negative change from baseline indicated improvement.
Time Frame: Baseline (Day 0) to Week 58
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 42
score on a scale
  Baseline | 2.3 (0.71)
  Change From Baseline to Week 58 | -1.6 (0.61)
Statistical Analysis 1: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference

8. Secondary Outcome: Mean Change From Baseline to Final Study Visit for Submental Skin Laxity Grade (SMSLG) Score
Description: The SMSLG scale integrated 3 skin features: skin wrinkling, adherence to underlying neck structures (bone and muscle), and redundancy (horizontal and vertical folds) assessed by the investigator using a 4-point scale where: 1=none, 2=mild, 3=moderate and 4=severe. A negative change from baseline indicated improvement.
Time Frame: Baseline (Day 0) to Week 58
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 42
score on a scale
  Baseline | 2.0 (0.62)
  Change From Baseline to Week 58 | -0.3 (0.62)
Statistical Analysis 1: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Test type: Other; p = 0.003, Paired t-test — P-value was based on paired t-test for the mean difference

9. Secondary Outcome: Mean Change From Baseline to Final Study Visit in Jawline Definition, Based on Independent Reviewer Assessment Using the ALJDS and Photographic Images
Description: The independent reviewer used photographic images collected at the time of the participant's live visit and the ALJDS to assess of loss of jawline definition using a 5-point scale where: 0=none, 1=mild, 2=moderate, 3=severe, 4=extreme. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 58
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
Number analyzed (Participants) | 42
score on a scale
  Both Side of the Face, Baseline | 2.9 (1.05)
  Both Side of the Face, End of Study | -0.7 (0.91)
  Right Side of the Face, Baseline | 2.7 (1.12)
  Right Side of the Face, End of study | -0.5 (0.98)
  Left Side of the Face, Baseline | 2.8 (1.08)
  Left Side of the Face, End of Study | -0.9 (0.98)
Statistical Analysis 1: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Both Side of the Face, End of Study; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference
Statistical Analysis 2: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Right Side of the Face, End of study; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference
Statistical Analysis 3: Comparison: BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine; Left Side of the Face, End of Study; Test type: Other; p < 0.001, Paired t-test — P-value was based on paired t-test for the mean difference

ADVERSE EVENTS:
Time Frame: Up to Week 58
Description: Safety Analysis Set included participants who are defined as Full Analysis Set (FAS) participants and those participants who underwent biopsy procedure but did not receive the BELKYRA® treatment.
Arm/Group | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 2/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine (N=53)
Volvulus (Gastrointestinal disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BELKYRA® and Juvéderm® VOLUMA™ With Lidocaine (N=53)
Nausea (Gastrointestinal disorders) | 6
Influenza like illness (General disorders) | 3
Injection site discolouration (General disorders) | 7
Injection site discomfort (General disorders) | 9
Injection site erythema (General disorders) | 11
Injection site hypoaesthesia (General disorders) | 29
Injection site induration (General disorders) | 24
Injection site mass (General disorders) | 31
Injection site pain (General disorders) | 39
Injection site pruritus (General disorders) | 5
Injection site reaction (General disorders) | 11
Injection site swelling (General disorders) | 39
Injection site warmth (General disorders) | 8
Swelling (General disorders) | 4
Injection site bruising (General disorders) | 38
Seasonal allergy (Immune system disorders) | 4
Lower respiratory tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 11
Weight decreased (Investigations) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Swelling face (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03425253/SAP_000.pdf
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03425253/Prot_001.pdf